CLINICAL TRIAL: NCT03142230
Title: Prevention of Pain Caused by the Oro-gastric Tube Laying in Neonatology
Acronym: DOLATSONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Sud Francilien (Other)
Collaborators: Centre National de Ressources de lutte contre la Douleur (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2015-A00427-42
Record Dates: First submitted 2017-03-28; First posted 2017-05-05 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Pain Score
Keywords: feeding tube; gastric; newborn infant; nursing; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized, multicentric, open-label, randomized study
Who Masked: Outcomes Assessor
Masking Description: The statistician is not aware of the control and experimental arms, called arms A and B in the results he must analyze.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-nutritive suction with holed baby bottle nipple (Experimental): A group using the holed baby bottle nipple
  Interventions: Other: the laying of the gastric tube and a group using the holed baby bottle nipple, the feeding tube ideally positioned at the center of the intersection pharyngeal
- Simple non-nutritive suction with personal pacifier (Active Comparator): A group using personal pacifier
  Interventions: Other: the laying of the gastric tube and a group with simple non-nutritive suction, the feeding tube passing next to the newborn's personal pacifier

INTERVENTIONS:
Other: the laying of the gastric tube and a group using the holed baby bottle nipple, the feeding tube ideally positioned at the center of the intersection pharyngeal — The newborn then receives the care with the introduction of the gastric tube after randomization with holed baby bottle nipple
  Arms: non-nutritive suction with holed baby bottle nipple
Other: the laying of the gastric tube and a group with simple non-nutritive suction, the feeding tube passing next to the newborn's personal pacifier — The newborn then receives the care with the introduction of the gastric tube after randomization with the newborn's personal pacifier
  Arms: Simple non-nutritive suction with personal pacifier

SUMMARY:
Subject of research : Evaluation of a technique of care to reduce the pain caused by the laying of the gastric tube in the newborn

DETAILED DESCRIPTION:
After inclusion, the nurse performs randomization by opening the envelope. The newborn then receives the care with the introduction of the gastric tube after randomization (experimental arm with holed baby bottle nipple and control arm: with pacifier). The treatment is filmed and recorded by a previously installed camera. The films are viewed by two independent experts from the pain of the study, to assess pain by scale score (DAN acute pain of the newborn

ELIGIBILITY:
Inclusion Criteria:

* Newborn term, or premature (from 32 weeks) from 48 hours to 14 days of life.
* Presence of sucking reflex
* Patient whose authors of parental authority have given their written consent for their participation
* Patient affiliated to or benefiting from a social security scheme

Exclusion Criteria:

* Newborn intubated or NIV and / or sedated
* Newborn with malformation (especially cleft palate)
* Contra-indication to sugar administration
* Newborn previously included in the study
* Administration of analgesics in the previous 8 hours
* Atresia of the unoperated esophagus
* Non-operated oeso-tracheal fistula
* Major swallowing disorders
* Necrotizing ulcerative colitis

Ages: 2 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
pain evaluation | Time of nurse care - thirty minutes maximum
  DAN SCALE

CONTACTS AND LOCATIONS:
Overall Officials: Michele Granier, MD, Study Director — Centre Hospitalier Sud Francilien
Locations (3):
- France (3):
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Centre Hospitalier de Saint-Denis, Saint-Denis

REFERENCES:
- [Derived] Darretain H, Laborne FX, Lagadec S, Garrigue B, Maillard F, Harbi F, Waszak P, Granier M, Galand N, Walter-Nicolet E, Razafimahefa H. An Analgesic Technique for Orogastric Tube Insertion in Newborns: DOLATSONG, a Randomized Multicentric Controlled Trial. J Perinat Neonatal Nurs. 2024 Oct-Dec 01;38(4):361-368. doi: 10.1097/JPN.0000000000000746. Epub 2024 Nov 7. PMID 38833575